CLINICAL TRIAL: NCT07167953
Title: MRI Technology for Greater Efficiency and Improved Value
Brief Title: The Spiral MRI Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-0948; 1R01EB036009-01A1 (NIH); A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); Protocol Version 6/2/2025 (Other: UW Madison)
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Brain MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Healthy Participants - Scan Efficiency (Experimental): Participants not otherwise undergoing a brain MRI
  Interventions: Device: Brain MRI - SOC and spiral
- Standard of Care (SOC) Brain MRI (Active Comparator): Participants undergoing SOC MRI
  Interventions: Device: Brain MRI
- Healthy Participants - Tau (Experimental): Participants not otherwise undergoing a brain MRI
  Interventions: Device: Brain MRI - spiral
- Healthy Participants - image quality (Experimental): Participants not otherwise undergoing a brain MRI
  Interventions: Device: Brain MRI - SOC and spiral
- Healthy Participants - SNR (Experimental): Participants not otherwise undergoing a brain MRI
  Interventions: Device: Brain MRI - spiral
- Healthy Participants - Gradient Derating (Experimental): Participants not otherwise undergoing a brain MRI
  Interventions: Device: Brain MRI - spiral

INTERVENTIONS:
Device: Brain MRI — 90 participants will undergo a 60 minute SOC brain MRI followed by 15 minute spiral MRI
  Arms: Standard of Care (SOC) Brain MRI
Device: Brain MRI - SOC and spiral — 6 participants will be scanned using 2 versions (SOC and spiral) pf 6 sequences (12 scans total).
  Arms: Healthy Participants - Scan Efficiency
Device: Brain MRI - spiral — 10 participants will be scanned with 3 sequences, 3 times (9 total scans per participants)
  Arms: Healthy Participants - Tau
Device: Brain MRI - SOC and spiral — 10 participants will be scanned using 2 versions (SOC and spiral) of 6 sequences (12 scans total).
  Arms: Healthy Participants - image quality
Device: Brain MRI - spiral — 10 participants will be scanned with 3 spiral sequences to achieve desired signal to noise ratio (SNR).
  Arms: Healthy Participants - SNR
Device: Brain MRI - spiral — 5 participants will be scanned with 2 pairs of 6 spiral sequences.
  Arms: Healthy Participants - Gradient Derating

SUMMARY:
The goal of this clinical trial is to find out if new Magnetic Resonance Imaging (MRI) computer software will:

* help make scans and exams faster
* reduce artifacts
* make MRI easier to understand
* allow technicians to focus more on the participant and less on the scanner

Participants will complete one brain MRI imaging session, lasting about 60 minutes.

DETAILED DESCRIPTION:
The overall goal of this application is to design technologies that improve the value of MRI, and specifically mitigate many of the complications that negatively impact this value. The scope of MRI value is vast, but can be expressed by efficiency (high patient throughput and consistent image quality), accessibility (better scope of use and equity of availability), safety, and user experience for the patient, technologist, and interpreting physician.

ELIGIBILITY:
Healthy Controls Inclusion Criteria:

* Adults at least 18 years
* Able to provide written informed consent on their own behalf

Brain MR Inclusion Criteria:

* Adults at least 18 years
* Able to provide written informed consent on their own behalf
* Scheduled for standard of care brain MRI

Exclusion Criteria (ALL):

* Unable or unwilling to provide informed consent
* Contraindication(s) to or inability to undergo MRI
* Currently pregnant
* Participants requiring intravenous (IV) conscious sedation for imaging are not eligible; participants requiring mild, oral anxiolytics for the clinical MRI will be allowed as long as the following criteria are met:
* participant has their own prescription for the medication
* informed consent process is conducted prior to the self-administration of the medication
* they come to the research visit with a driver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2028-08 (Estimated); Primary Completion 2031-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Image quality - decreasing scan time | 60 minutes
  Participants will be scanned using 2 versions (standard and spiral) of 6 sequences (12 scans total). For each sequence pair, scan time will be sped up. Image quality will be compared between the 2 versions.
Image quality - tau | 60 minutes
  Measuring whether image quality is sufficient for routine diagnostic interpretation - specifically robustness to artifacts. The independent variable is a scanning parameter called tau, which researchers want to be long (because it makes the total scan time shorter). Researchers will compare the value of tau between SOC imaging and spiral. They will use a 5-point Likert scale to compare, where 1= undiagnostic (unacceptable), 2 = spiral scans slightly worse than SOC but acceptable, 3= spiral scans same as SOC (acceptable), 4= spiral scans slightly better than SOC (acceptable), 5=spiral scans much better than SOC (acceptable).
Image quality - consistent scan time | 60 minutes
  Participants will be scanned using 2 versions (standard and designed) of 6 sequences (12 scans total). Scan time will remain the same for each pair. Radiologists will compare each pair for differences in image quality using a 5-point Likert scale where 1= A much worse than B, 2=A slightly worse than B, 3=A comparable to B, 4=A slightly better than B, 5=A much better than B. A=new spiral scans and B=SOC scans.
Signal to Noise Ratio (SNR) | 60 minutes
  Measuring the SNR in images, by measuring the signal strength in the image and the calculated noise in those images and taking the ratio. Researchers will compare this SNR to that which their methods predicted.
Image quality - acoustic comfort | 60 minutes
  Image quality will be compared between running at full strength, which is noisy, and running at reduced strength, which should be quieter. A 5-point Likert scale will be used, where 1= A much worse than B, 2=A slightly worse than B, 3=A comparable to B, 4=A slightly better than B, 5=A much better than B. A=spiral scans with full gradient strength and B=spiral scans with reduced gradient strength (that should be quieter).
Acoustic noise | 60 minutes
  Scans will be compared between running at full strength and running at reduced strength. Participants will rate the acoustic noise using a 5-point Likert scale, where 1= A much louder than B, 2=A slightly louder than B, 3=A comparable to B, 4=A slightly quieter than B, 5=A much quieter than B. A=spiral scans with full gradient strength and B=spiral scans with reduced gradient strength.
Difference in Image quality | 60 minutes
  Based on the results of the other 5 outcome measures, specifically whether scan time impacts image quality, the desired time will be used and scans will be compared between SOC and their method. Image quality will be measured using a 5-point Likert scale, where 1= A much worse than B, 2=A slightly worse than B, 3=A comparable to B, 4=A slightly better than B, 5=A much better than B. A=new spiral scans and B=SOC scans.

CONTACTS AND LOCATIONS:
Overall Officials: James Pipe, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States